CLINICAL TRIAL: NCT02583880
Title: Screening Day Latin America to Assess Disease-related Malnutrition and Clinical Nutrition Practice in ICU Patients
Brief Title: Screening Day Latin America
Status: Completed | Type: Observational
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Other Study IDs: NScr-001-CNI
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-09

CONDITIONS: Nutritional Status; Malnutrition; Caloric Deficit
Keywords: nutritional status; malnutrition; energy intake; caloric deficit; ICU; hospital; enteral nutrition; parenteral nutrition; nutrition
MeSH Terms: conditions — Malnutrition; Hyperphagia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a survey which will be performed on a specific day (the "Screening Day") in Latin American ICUs.

In eligible patients who receive enteral or parenteral nutrition a retrospective calculation of the "caloric deficit" will be performed. The caloric deficit is the difference between energy target of each patient and actually administered calories.

DETAILED DESCRIPTION:
The Screening Day Latin America is a non-interventional, cross-sectional and retrospective study. The study focusses on patients receiving enteral (tube feeding, EN) and/or parenteral nutrition (PN).

All patients hospitalized on the defined Screening Day in participating ICUs will be checked for eligibility. In eligible patients the patient charts will be reviewed and the following parameters will be documented:

* Caloric deficit (daily target energy - actually administered energy via EN and PN). The caloric deficit will be calculated for 1 to up to 5 days before the Screening Day. The analysis will be done for each day and for the complete documentation period up to 5 days. Primary focus will be the caloric deficit on Day -1.
* Nutritional status of the patient based on information from the patient charts. For this, three tools will be applied independently: Subjective Global Assessment (SGA), NUTRIC Score, ESPEN diagnosis of malnutrition

The study will be performed in 8 Latin American countries.

Data will be recorded anonymously in an electronic case report form.

The study data of this explorative study will be analyzed using descriptive statistical methods.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if the following criteria are fulfilled:

* Critically ill adult (≥18 years of age) patients, including critically ill major gastrointestinal surgery patients
* Patient is hospitalized in Intensive Care Unit (ICU) on the Screening Day
* Patients receiving enteral nutrition (EN; tube feeding only) and/or parenteral nutrition (PN) on the Screening Day and the day before the Screening Day
* Initiation of enteral nutrition (EN) and/or parenteral nutrition (PN) during ICU admission and at least one day before the Screening Day

A critically ill patient is defined as a patient with at least one organ failure.

Exclusion Criteria:

The following patients are excluded from the documentation:

* Critically ill burn patients
* Patients on the Intensive Care Unit (ICU) for surveillance without needing enteral nutrition (EN) and/or parenteral nutrition (PN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients receiving enteral and/or parenteral nutrition, hospitalized in the Intensive Care Units (ICUs) of the participating hospitals on the Screening Day
Sampling Method: Non-Probability Sample
Enrollment: 1162 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Caloric deficit on the day before the Screening Day | On the day before the Screening Day (day -1)
  The caloric deficit on the day before the Screening Day will be derived by subtracting the provided calories from EN, PN and additional sources of caloric intake (e.g., dextrose-containing solutions, propofol emulsion) from the defined caloric target.
  Equation: Caloric Deficit = Target Calories - Given Calories
  If a caloric target is not provided/defined it will be assumed to be:
  * 20 kcal/kg/day actual body weight for the first 6 days after ICU admission
  * 25 kcal/kg/day actual body weight after day 6 of ICU admission period

SECONDARY OUTCOMES:
Cumulative caloric deficit on days -1 to -5 before the screening day | Days -1 to -5
  The cumulative caloric deficit is the sum of the caloric deficit on day -1 + caloric deficit on Day -2 + caloric deficit on Day -3 + caloric deficit on Day -4 + caloric deficit on Day -5, depending on the number of days on the ICU
Nutritional status of the patient | The Screening Day (Day 0) and the day of admission to the Intensive Care Unit (ICU)
  The nutritional status is assessed by using three different tools independently: The Subjective Global Assessment (SGA), the NUTRIC Score, and the ESPEN diagnosis of malnutrition
Current use of enteral and parenteral nutrition | At Screening Day
  The type and volume of administered enteral and parenteral nutrition will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: John F Stover, MD, Study Chair — Fresenius Kabi Deutschland GmbH, Borkenberg 14, 61440 Oberursel, Germany
Locations (121):
- Argentina (19):
  - Fumeba, Bahía Blanca, Buenos Aires
  - Hospital Penna, Bahía Blanca, Buenos Aires
  - UAI, Buenos Aires, Buenos Aires
  - Hospital Británico, Caba, Buenos Aires
  - Hospital Carrillo, Ciudadela, Buenos Aires
  - Hospital Fernandez, Caba, Buenos Aires F.D.
  - Sanatorio San Jose, Caba, Buenos Aires F.D.
  - Sanatorio Colegiales, Caba, Buenos Aires F.D.
  - Hospital Raul Ferreyra, Córdoba, Córdoba Province
  - Sanatorio Allende, Córdoba, Córdoba Province
  - Hospital San Martín, La Plata, GBA
  - Hospital El Cruce, San Juan Bautista, GBA
  - Hospital Pablo Soria, San Salvador de Jujuy, Jujuy Province
  - Sanatorio Norte, San Salvador de Jujuy, Jujuy Province
  - CMIC, Neuquén, Neuquén Province
  - Hospital Eva Perón, Granadero Baigorria, Rosario
  - Hospital Oñativia, Salta, Salta Province
  - Hospital Cullen, Santa Fe, Santa Fe Province
  - H. Centro de Salud, San Miguel de Tucumán, Tucumán Province
- Brazil (13):
  - Irmandade Nossa Senhora Das Merces, Montes Claros, Minas Gerais
  - Hospital Das Clinicas Minas Gerais, Belo Horizonte
  - Hospital Felicio Rocho, Belo Horizonte
  - Hosp de Caridade São Vicente de Paulo, Jundiaí
  - Antonio Pedro (Huap), Niterói
  - Quinta D'Or, Rio de Janeiro
  - Santa Casa de Misericórdia Da Bahia (Hosp St Izabel), Salvador
  - Hospital Beneficência Portuguesa de Sp, São Paulo
  - Hospital Das Clinicas São Paulo, São Paulo
  - Hospital Sirio Libanes, São Paulo
  - Hospital Sta Marcelina de Itaquera, São Paulo
  - Instituto de Assistência Médica Ao Servidor Público Estadual - Iamspe, São Paulo
  - Hospital Metropolitano, Serra
- Chile (22):
  - Hospital Regional de Antofagasta, Antofagasta, Antofagasta
  - Hospital Dr. Gustavo Fricke, Viña del Mar, Región de Valparaíso
  - Hospital las Higueras, Concepción, Región del Biobío
  - Salvador, Providencia, Santiago Metropolitan
  - Clínica Dávila, Santiago, Santiago Metropolitan
  - Hospital Luis Tisne, Santiago, Santiago Metropolitan
  - Hospital San Jose, Santiago, Santiago Metropolitan
  - Hospital Universidad Católica, Santiago, Santiago Metropolitan
  - Indisa, Santiago, Santiago Metropolitan
  - San Borja, Santiago, Santiago Metropolitan
  - San Juan de Dios, Santiago, Santiago Metropolitan
  - Hospital Clínico Regional de Concepcion Grant Benavente, Concepción
  - Hospital Militar de Santiago, La Reina
  - Clínica Bicentenario, Región Metropolitana
  - Hospital Clínico de la Universidad de Chile, Región Metropolitana
  - Hospital Barros Luco-Trudeau, Santiago
  - Hospital Clínico La Florida, Santiago
  - Hospital Dipreca, Santiago
  - Mutual de Seguridad, Santiago
  - Hospital de Talca, Talca
  - Hospital Dr. Hernán Henríquez Aravena, Temuco
  - Hospital Naval, Viña del Mar
- Colombia (22):
  - Clínica de la Costa, Barranquilla, Atlántico
  - Hospital del Cari, Barranquilla, Atlántico
  - Clínica Universitaria Colombia, Bogotá, Bogota D.C.
  - Hospital El Tunal, Bogotá, Bogota D.C.
  - Hospital San José Sociedad de Cirugía de Bogotá, Bogotá, Bogota D.C.
  - Hospital Universitario Clínica San Rafael, Bogotá, Bogota D.C.
  - Hospital Universitario Mayor MEDERI, Bogotá, Bogota D.C.
  - Hospital San José de Popayán, Popayán, Cauca Department
  - Clínica Evaluamos, Montería, Departamento de Córdoba
  - IMAT, Montería, Departamento de Córdoba
  - Clinica San José de Cúcuta, Cúcuta, Norte de Santander Department
  - FOSCAL, Floridablanca, Santander Department
  - Clínica Rey David, Cali, Valle del Cauca Department
  - Fundación Valle de Lili, Cali
  - Clínica Unipamplona, Cúcuta
  - Hospital Erasmo Meoz, Cúcuta
  - FOSUNAB, Floridablanca
  - SES Hospital de Caldas, Manizales
  - Clínica Medellín, Medellín
  - Fundación Hospitalaria San Vicente de Paul, Medellín
  - Hospital General de Medellín, Medellín
  - Promotora Clínica Las Américas, Medellín
- Ecuador (14):
  - Hospital Carrasco Arteaga, Cuenca
  - Hospital Vicente Corral, Cuenca
  - Hospital Clínica Kennedy, Guayaquil
  - Hospital IESS Teodoro Maldonado Carbo, Guayaquil
  - Hospital Luis Vernaza, Guayaquil
  - Hospital Universitario, Guayaquil
  - Hospital de las Fuerzas Armadas, Quito
  - Hospital Carlos Andrade Marin, Quito
  - Hospital de la Policia, Quito
  - Hospital de los Valles, Quito
  - Hospital Eugenio Espejo, Quito
  - Hospital IESS San Francisco, Quito
  - Hospital Inglés, Quito
  - Hospital Metropolitano, Quito
- Mexico (15):
  - Centro Médico Chiapas Nos Une "Dr. Jesús Gilberto Goméz Maza", Tuxtla Gutiérrez, Chiapas
  - Central Universitario, Chihuahua City, Chihuahua
  - General de Cd. Juarez, Ciudad Juárez, Chihuahua
  - Hospital General de Tijuana, Tijuana, Estado de Baja California
  - Hospital General Pachuca, Pachuca, Hidalgo
  - Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Hospital General Balbuena, Mexico City, Mexico City
  - Hospital General de México, Mexico City, Mexico City
  - Centro Médico Dalinde, Mexico City, Mexico City
  - Hospital Universitario, Monterrey, Nuevo Léon
  - Hospital Metropolitano, San Nicolás de los Garza, Nuevo Léon
  - Isem Centro Médico, Toluca, State of Mexico
  - Hospital Regional de Veracruz, Veracruz, Veracruz
  - CEMEV, Xalapa, Veracruz
  - Hospital de la Soledad, San Luis Potosí City
- Caja del Seguro Social, Panama City, Panama
- Peru (15):
  - Hospital Hipolito Unanue, El Agustino, Lima region
  - Hospital Guillermo Kaelin de la Fuente, Lima, Provincia de Líma
  - Centro Médico Naval, Callao
  - Hospital Alberto Leopoldo Barton Thompson, Callao
  - Hospital Alberto Sabogal Sologuren, Callao
  - Hospital Regional Trujillo, La Libertad
  - Clinica Centenario, Lima
  - Clínica Adventista Good Hope, Lima
  - Hospital 2 de Mayo, Lima
  - Hospital Edgardo Rebagliati Martins, Lima
  - Hospital Guillermo Almenara Irigoyen, Lima
  - Hospital Luis Saenz de la Policia, Lima
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Santa Rosa, Lima
  - Hospital Víctor Lazarte de Red Asistencial La Libertad de EsSalud, Trujillo La Libertad